CLINICAL TRIAL: NCT06575140
Title: Pilot Randomized Controlled Trial Assessing Associative Peripheral Stimulation (APS) for Reduction of Motor Impairment During Acute Period of Stroke Recovery
Brief Title: Associative Peripheral Stimulation for Reduction of Motor Impairment During Acute Period of Stroke Recovery
Acronym: APS-PILOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed A. Rahim (Other)
Responsible Party: Sponsor-Investigator, Ahmed A. Rahim, Sponsor-Investigator, APS Trial Group
Organization: APS Trial Group (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APS-PILOT
Record Dates: First submitted 2019-03-24; First posted 2024-08-28 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Stroke; Stroke, Acute; Stroke, Ischemic; Stroke, Hemorrhagic; Hemiparesis; Hemiparesis;Poststroke/CVA; Weakness of Extremities as Sequela of Stroke; Stroke Sequelae; Upper Extremity Paresis
Keywords: Stroke Rehabilitation; Associative Peripheral Stimulation
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke; Paresis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Group A (Experimental): Treatment
  Interventions: Device: Associative Peripheral Stimulation (APS) 1.0
- Group B (Active Comparator): Control
  Interventions: Device: Peripheral Neuromuscular Stimulation

INTERVENTIONS:
Device: Associative Peripheral Stimulation (APS) 1.0 — Associative peripheral stimulation paired with rehabilitative exercises.
  Arms: Group A
Device: Peripheral Neuromuscular Stimulation — Random peripheral stimulation paired with rehabilitative exercises.
  Arms: Group B

SUMMARY:
Associative Peripheral Stimulation (APS) is a non-invasive therapy intended for stroke rehabilitation involving transcutaneous electrical muscle stimulation paired with voluntary movement. This pilot study investigates whether APS applied during the acute phase of stroke recovery may reduce impairment and improve function in the affected upper extremity.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed ischemic or hemorrhagic stroke no earlier than 7 days prior to enrollment;
2. Presentation of hemiparesis or paralysis of the upper extremity due to stroke;
3. Ability to comprehend and follow study instructions;
4. Ability to initiate finger extension (≥3°) at least three times per minute;
5. Fugl-Meyer Assessment (Upper Extremity) score of <47.

Exclusion Criteria:

1. Contraindications, intolerance, or high sensitivity to the experimental protocol;
2. History of upper-extremity disability prior to the index stroke;
3. Neurological conditions (other than stroke) affecting motor function;
4. Treatment of spasticity/increased tone in the affected upper extremity (e.g., with Botox injection);
5. Lack of access to a safe and suitable place of discharge for experimental sessions and follow-up visits.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-18 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Average of Range of Motion (ROM) | 5 weeks
  Measure of distal extensor function (wrist and fingers). Unit of measurement: degrees (°). Higher scores indicate better outcomes.
Fugl-Meyer Assessment Upper-Extremity (FMA-UE) | 5 weeks
  Measure of motor recovery in stroke patients with hemiparesis. Scoring range: 0 to 66. Higher scores indicate better outcomes.

SECONDARY OUTCOMES:
Maximum Average of Range of Motion (ROM) | 3 months
  Measure of distal extensor function (wrist and fingers). Unit of measurement: degrees (°). Higher scores indicate better outcomes.
Fugl-Meyer Assessment Upper-Extremity (FMA-UE) | 3 months
  Measure of motor recovery in stroke patients with hemiparesis. Scoring range: 0 to 66. Higher scores indicate better outcomes.
Action Research Arm Test (ARAT) | 5 weeks
  Measure of four functional domains: grasp, grip, pinch, and gross arm movement. Scoring Range: 0 to 57. Higher scores indicate better outcomes.
Action Research Arm Test (ARAT) | 3 months
  Measure of four functional domains: grasp, grip, pinch, and gross arm movement. Scoring Range: 0 to 57. Higher scores indicate better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel San Juan Orta, MD, Study Director — National Institute of Neurology & Neurosurgery
Locations (3):
- Mexico (3):
  - General Hospital of Mexico, Mexico City
  - La Raza National Medical Center, Mexico City
  - National Institute of Neurology & Neurosurgery, Mexico City

IPD SHARING:
Plan to Share IPD: No
Individual participant data shall not be made available to other researchers.